CLINICAL TRIAL: NCT03388541
Title: Does LOW Dose DEXmedetomidine After Cardiopulmonary Bypass Separation Decrease the Incidence of DELirium: A Double-blind Randomized Placebo-controlled Study (LOWDEXDEL Study)
Brief Title: Low Dose Dexmedetomidine and Delirium After Cardiac Surgery
Acronym: LOWDEXDEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Mona Momeni, MD, PhD, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/24JUL/374
Record Dates: First submitted 2017-08-01; First posted 2018-01-03 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Cardiac Surgical Procedures
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine will be administered at 0.4ug/kg/h (5mL/h) starting at the closure of the chest and continued during 10h.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): NaCl 0.9% will be administered at 5mL/h starting at the closure of the chest and continued during 10h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be started at 5mL/h while the patient is still in the operating room. The patient will be transferred to the intensive care unit with a sedative regimen based on propofol.
  Arms: Dexmedetomidine
Drug: Placebo — A continuous infusion of NaCL 0.9% will be started at 5mL/h while the patient is still in the operating room. The patient will be transferred to the intensive care unit with a sedative regimen based on propofol.
  Arms: Placebo

SUMMARY:
Delirium after cardiac surgery can occur in up to 50% of the patients and has been shown to be significantly associated with increased morbidity and mortality. Advanced age is a significant risk factor of delirium.

Numerous studies have shown that sedation with high doses of Dexmedetomidine in the ICU reduces the incidence of postoperative delirium. On the other hand animal studies have shown neuroprotective effects of Dexmedetomidine by means of stimulating alpha2A-adrenoceptors.

It is not clear whether the administration of a low dose Dexmedetomidine in cardiac surgery would have any neuroprotective effects by stimulating the alpha 2A-receptors and as such would decrease the incidence of postoperative delirium.

DETAILED DESCRIPTION:
Postoperative delirium (PD) is a common problem in cardiac surgical patients. Its incidence varies among studies and can reach up to 50% of the patients. PD is associated with increased morbidity and mortality. Its occurrence is the resultant between the predisposing factors and the precipitating factors. Age seems to be a significant predisposing factor. In this regard the pathophysiology of PD is not yet fully understood. There are several hypothetical mechanisms for the development of PD. The first hypothesis is cerebral ischemia and BBB breakdown. The second hypothesis is neuro-inflammation. Peripheral pro-inflammatory mediators especially released during surgery would interact with the brain. Otherwise there is the problem of sleep deprivation/fragmentation in patients admitted to the hospital.

Dexmedetomidine is a potent and more selective alpha2-adrenergic receptor than clonidine. Studies have demonstrated that it has neuroprotective and anti-inflammatory actions.

Numerous studies including trials in cardiac surgery have shown a decreased incidence of delirium when Dexmedetomidine was used as sedative in the ICU compared with other sedatives acting on the GABA receptors. However, in these studies high doses of Dexmedetomidine were used for periods up to 24h. Dexmedetomidine was started in the ICU and was not compared in a double-blind fashion with placebo. In a recent randomized double-blind placebo-controlled trial a very low dose of Dexmedetomidine decreased the occurrence of PD when compared to placebo. However this study was performed in non-cardiac patients. Moreover the patients were included after their arrival in the ICU, which means that those patients who were intubated at their arrival in the ICU were not included. And again the study medication was only started after arrival in the ICU.

The aim of this study is to elucidate whether the administration of Dexmedetomidine at a low dose would decrease the incidence of PD in elderly patients undergoing cardiac surgery. The hypothesis is that Dexmedetomidine at low doses, by only stimulating the alpha2A adrenoceptors,would have neuroprotective affects ans as such decrease the incidence of PD. Dexmedetomidine would also have anti-inflammatory effects and effects on the quality of sleep. Both mechanisms would play a role in the pathophysiology of PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Hepatic dysfunction (hepatic function tests 3 times the normal value)
* Preoperative renal replacement therapy
* Preoperative delirium
* Emergency surgery not allowing neurologic evaluation by MMSE
* Mini invasive cardiac surgery
* Patients not speaking French

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
The incidence of delirium | Through study completion, an average of 30 days
  The incidence of delirium detected by means of CAM-ICU and CAM

SECONDARY OUTCOMES:
Number of days spent in delirium | Through study completion, an average of 30 days
  Total number of days in a delirious state
ICU stay | Through study completion, an average of 30 days
  The duration of days admitted in the ICU and in the hospital
Total dose of analgesics | Through study completion, an average of 30 days
  Total dose of analgesics used in the ICU
Total dose of vasopressors | Through study completion, an average of 30 days
  Total dose of vasopressors used in the ICU
Pace maker necessitation | Through study completion, an average of 30 days
  Number of patients needing external pacing
Hospital stay | Through study completion, an average of 30 days
  The duration of days admitted in the hospital
Total dose sedatives | Through study completion, an average of 30 days
  Total dose of sedatives used in the ICU
Total dose of inotropic agents | Through study completion, an average of 30 days
  Total dose of inotropic agents used in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Mona Momeni, MD,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paris A, Mantz J, Tonner PH, Hein L, Brede M, Gressens P. The effects of dexmedetomidine on perinatal excitotoxic brain injury are mediated by the alpha2A-adrenoceptor subtype. Anesth Analg. 2006 Feb;102(2):456-61. doi: 10.1213/01.ane.0000194301.79118.e9. PMID 16428542
- [Background] Maier C, Steinberg GK, Sun GH, Zhi GT, Maze M. Neuroprotection by the alpha 2-adrenoreceptor agonist dexmedetomidine in a focal model of cerebral ischemia. Anesthesiology. 1993 Aug;79(2):306-12. doi: 10.1097/00000542-199308000-00016. PMID 8102042
- [Background] Jiang L, Hu M, Lu Y, Cao Y, Chang Y, Dai Z. The protective effects of dexmedetomidine on ischemic brain injury: A meta-analysis. J Clin Anesth. 2017 Aug;40:25-32. doi: 10.1016/j.jclinane.2017.04.003. Epub 2017 Apr 17. PMID 28625441
- [Background] Tasdogan M, Memis D, Sut N, Yuksel M. Results of a pilot study on the effects of propofol and dexmedetomidine on inflammatory responses and intraabdominal pressure in severe sepsis. J Clin Anesth. 2009 Sep;21(6):394-400. doi: 10.1016/j.jclinane.2008.10.010. PMID 19833271
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Shehabi Y, Grant P, Wolfenden H, Hammond N, Bass F, Campbell M, Chen J. Prevalence of delirium with dexmedetomidine compared with morphine based therapy after cardiac surgery: a randomized controlled trial (DEXmedetomidine COmpared to Morphine-DEXCOM Study). Anesthesiology. 2009 Nov;111(5):1075-84. doi: 10.1097/ALN.0b013e3181b6a783. PMID 19786862
- [Background] Djaiani G, Silverton N, Fedorko L, Carroll J, Styra R, Rao V, Katznelson R. Dexmedetomidine versus Propofol Sedation Reduces Delirium after Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2016 Feb;124(2):362-8. doi: 10.1097/ALN.0000000000000951. PMID 26575144
- [Derived] Momeni M, Khalifa C, Lemaire G, Watremez C, Tircoveanu R, Van Dyck M, Kahn D, Rosal Martins M, Mastrobuoni S, De Kerchove L, Zango SH, Jacquet LM. Propofol plus low-dose dexmedetomidine infusion and postoperative delirium in older patients undergoing cardiac surgery. Br J Anaesth. 2021 Mar;126(3):665-673. doi: 10.1016/j.bja.2020.10.041. Epub 2020 Dec 24. PMID 33358336